CLINICAL TRIAL: NCT06297447
Title: Keeping It Simple Study (KISS) - Pain Science Education for Patients With Chronic Musculoskeletal Pain Undergoing Community-based Rehabilitation: A Multicenter Randomized Controlled Trial
Brief Title: Keeping it Simple Study (KISS)
Acronym: KISS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bettina Eiger (Other)
Collaborators: University of Southern Denmark (Other); Aalborg University (Other); Central Denmark Region (Other); Vrije Universiteit Brussel (Other)
Responsible Party: Sponsor-Investigator, Bettina Eiger, Principal Investigator, Aalborg University
Organization: Aalborg University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: N-20230073
Record Dates: First submitted 2024-02-29; First posted 2024-03-07 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Musculoskeletal Pain; Chronic Pain
Keywords: Pain education; Musculoskeletal Pain; Chronic pain; PNE4Adults; Adults; Rehabilitation; Health literacy
MeSH Terms: conditions — Musculoskeletal Pain; Chronic Pain

STUDY DESIGN:
Intervention Model Description: Multicenter randomized controlled, superiority trial with a 2-group parallel design.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Randomization will be stratified by cite. Block randomization in random concealed block sizes of 4 to 6 (1:1) into two parallel groups is used to avoid imbalance in the randomization between intervention groups. A person not otherwise affiliated with the study will generate the randomization sequence.The randomization will be coded (Group 1 or 2), thus the primary investigator (BE) will not know the code to the groups.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- "Usual care" (Active Comparator): "Usual Care": The control group receives unrestricted "usual care". It could include a patient interview with individual goal setting and subsequent rehabilitation using cardio and strengthening exercises towards achieving the determined goals. It will be delivered by an authorized physiotherapist, and the intervention is determined by patient preferences, physiotherapist's clinical reasoning, and available resources.
  Interventions: Other: Usual care
- PNE4Adults - pain science education (Experimental): PNE4Adults: In this group, the participants will receive an add-on individualized PSE in addition to the usual care with the PNE4Adults resource. The PNE4Adults session will follow the developed manual (http://www.paininmotion.be/pne4kids) and will be delivered by a physiotherapist in two sessions of each 30-45 minutes, shortly following the first meeting. Firstly, the function of a normal pain system is introduced, with examples of the pain being overly or under protective. Then, the patient teaches back giving the therapist the opportunity to evaluate the understanding and, if necessary, repeat essential key messages. Secondly, the sensitized pain system is explained. Thirdly, the subject is asked to reflect on this new information in relation to his/her own situation. Subsequently, the new knowledge is integrated in "usual care" with any additional measures that need to be included, e.g., graded exposure, stress relief, graded activity, and cognitive therapies.
  Interventions: Other: PNE4Adults - pain science education

INTERVENTIONS:
Other: PNE4Adults - pain science education — Is formerly described under arm descriptions
  Arms: PNE4Adults - pain science education
Other: Usual care — Is formerly described under arm descriptions
  Arms: "Usual care"

SUMMARY:
Problem: The number of patients living with chronic musculoskeletal (MSK) pain has steadily increased over the past decade with costs rising equally. Long-standing pain is associated with significant maladaptive beliefs about pain, psychological characteristics and associated behaviors which involve structural and functional neurobiological characteristics which share common pathophysiological mechanisms as chronic pain. The investigators recent priority setting partnership investigated the research priorities from 1000 patients with chronic MSK pain, relatives, and clinicians. Better pain education was rated as one of the three most important research areas.

Solution: Pain science education has the potential to target maladaptive psychological and behavioral components that may contribute to the maintenance of chronic pain. The KISS project will evaluate the effect of a pain neuroscience education program (PNE4Adults) on rehabilitation outcomes in patients with chronic MSK pain. This intervention has the potential to change beliefs and behaviors surrounding pain in patients with chronic MSK pain. If this is successful in disrupting maladaptive cycles contributing to chronicity, this may improve outcomes for many thousand citizens.

DETAILED DESCRIPTION:
Introduction: Between 20% and 33% of people across the globe live with a painful musculoskeletal (MSK) condition. Costs correspond to almost 2% of the gross domestic products of European countries, posing a challenge for health care systems across the world. Patients with chronic musculoskeletal pain have a high use of healthcare, reduced work ability, loss of productivity, and loss of quality of life. Current care guidelines underline that pain science education (PSE) is a vital part of the care delivered to people suffering from chronic pain. PSE is thought in part to attenuate central sensitization and improve self-efficacy potentially mediated through decreased pain catastrophizing and modulating nocebo-related effects. On a patient level, PSE has been shown to reduce pain catastrophizing, pain intensity, and fear-avoidance in addition to improved physical functioning, self-efficacy, and pain knowledge. Combining exercise and PSE shows greater short-term improvements in pain, disability, kinesiophobia, and pain catastrophizing compared to exercise alone and the RESTORE-trial showed the benefit of adding cognitive components. On a societal level, PSE has further shown to minimize health expenses. However, some of the proposed barriers include training of the therapist delivering the education, access to training material, time during consultation, and patients' health literacy levels. Even in Denmark, a country with a highly educated population, the prevalence of people with inadequate health literacy is high, with nearly 4 out of 10 people facing difficulties accessing, understanding, appraising, and applying health information. This underlines the need to consider novel ways of delivering PSE across all levels of health literacy.

Due to the lack of tools to facilitate PSE programs, the investigators adapted an existing pain science education program that was developed by Pas et al. (2018) (PNE4Kids) to teach children with chronic pain about the underlying biopsychosocial mechanisms contributing to pain. The adapted version, named PNE4Adults, consists of a manual for the therapist and a board game to enhance engagement and participant involvement. It provides the therapist with a clear "how-to" manual and an accessible way for patients to understand the complex concept of pain. This new PSE program may also hold promise for adult patients with low levels of health literacy and enhance learning due to its practical tools and build-in teach-back. The focus on integrating PSE into rehabilitation may enhance the therapeutic alliance needed to facilitate the patients' ability to manage their own symptoms. The investigators feasibility study in adult patients with chronic MSK pain in community-based rehabilitation (Eiger, Rathleff et al. 2024 - under review) showed that PNE4Adults was well accepted (100%) and understandable by all (100%) patients, including those with low levels of health literacy. Qualitive interviews revealed that patients (irrespective of their health literacy) acquired a deeper understanding of their own situation and their pain. This novel approach may reduce the inequality in delivering of pain education.

Purpose of Sub-project 1 The primary aim of the KISS-project is to evaluate the added effect of PSE ('PNE4Adults') to "usual care" compared to "usual care" alone in community-based rehabilitation.

The investigators hypothesis is PSE plus "usual care" will result in a larger improvement of musculoskeletal health (MSK-HQ) after 3 months (primary endpoint) compared to patients undergoing "usual care" in the municipality.

Purpose of Sub-project 2 The secondary aim is to use a process evaluation to understand how it works, and for whom the program works.

The purpose of the process evaluation is to understand how it worked and for whom, and not if it worked. The investigators will combine in-house registrations from the municipality, clinician observations, individual interviews, and focus-group interviews to answer what works for whom and under which circumstances. This will give the investigators additional insights into the novel PSE intervention, shedding light on how it induces change and uncovering any potential unintended consequences. This will support future implementation pending results.

ELIGIBILITY:
Inclusion Criteria:

* Patients referred for rehabilitation in the municipalities Køge, Holbæk, and Solrød
* With chronic (>3 months) musculoskeletal pain.
* Adult patients (≥18 years) - no upper limit
* Able to understand, speak, and write Danish.

Exclusion Criteria:

* Known cognitive deficits (e.g., dementia).
* Diagnosed with cancer or other serious pathologies, e.g., cauda equina.
* Pregnancy
* Drug addiction defined as the use of cannabis, opioids, or other drugs.
* Neurologic or psychiatric diagnoses that hinder participation, e.g., stroke and borderline.
* Lack of ability to cooperate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-03-11 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Musculoskeletal Health Questionnaire (MSK-HQ) | Primary endpoint at 3 months, additional at 6 weeks and 6 months
  Musculoskeletal (MSK) Health assessed by the Musculoskeletal Health Questionnaire. Score from 0 to 56. Higher scores reflect better MSK health, and better outcome

SECONDARY OUTCOMES:
Mean Pain intensity | At 6 weeks, 3 months and 6 months
  Average of two numeric rating scales (most severe pain and average pain past 24 hours). Scores from 0 to 10. Higher scores reflect more intense pain, and worse outcome.
Pain interference | At 6 weeks, 3 months and 6 months
  Pain interference subscale of Brief Pain Inventory, Score from 0 to 70, higher scores reflect more bothersome and worse outcomes.
Concept of pain | At 6 weeks, 3 months and 6 months
  Measured on the Adult Concept of Pain Inventory, Danish. Scores from 0 to 52. Higher scores reflect more alignment with contemporary pain science knowledge and better outcome.
Pain catastrophizing | At 6 weeks, 3 months and 6 months
  Measured on the Pain Catastrophizing Scale, Score from 0 to 52. Higher scores reflect worse outcomes
Fear of movement | At 6 weeks, 3 months and 6 months
  Measured on the Tampa Scale of Kinesiophobia (TSK-11), scores between 11 and 44. Higher scores reflect more fear of movement and worse outcomes
Patient specific functional limitation | At 6 weeks, 3 months and 6 months
  Patient-Specific Functional Scale, scores from 0 to 10. Higher scores reflect better outcomes
Patient impression of change | At 6 weeks, 3 months and 6 months
  Global Impression of Change Scale (GISC), From "very much improved" to "very much worse".
Patient satisfaction with current symptom state | At 6 weeks, 3 months and 6 months
  Measured with the Patient Acceptable Symptom State (PASS), Yes/No answer. No is worse outcome.
Pain Self-efficacy | At 6 weeks, 3 months and 6 months
  Pain Self-efficacy Questionnaire (PSEQ), scores from 0 to 60, higher scores reflect higher self-efficacy and better outcome.
Adverse events | "through study completion, an average of 6 months".
  Any adverse events will be noted. The higher the number, the worse outcome

CONTACTS AND LOCATIONS:
Overall Officials: Bettina Eiger, PhD-student, Principal Investigator — Aalborg University
Locations (3):
- Denmark (3):
  - Træningsenheden, Holbæk Municipality, Holbæk, Region Sjælland
  - Træningsenheden, Køge Municipality, Køge, Region Sjælland
  - Genoptræningscenteret, Solrød Municipality, Solrød Strand, Region Sjælland

DOCUMENTS (2):
  • Study Protocol (2024-03-06): https://cdn.clinicaltrials.gov/large-docs/47/NCT06297447/Prot_000.pdf
  • Statistical Analysis Plan (2024-12-20): https://cdn.clinicaltrials.gov/large-docs/47/NCT06297447/SAP_001.pdf